CLINICAL TRIAL: NCT00136773
Title: Effects of Amlodipine/Benazepril on Albuminuria in Hypertensive Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCIB002FUS12
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2008-03

CONDITIONS: Albuminuria
Keywords: Albuminuria; Type 2 diabetes mellitus; Hypertension
MeSH Terms: conditions — Albuminuria; Diabetes Mellitus, Type 2; Hypertension | interventions — benazepril

INTERVENTIONS:
Drug: amlodipine/benazepril

SUMMARY:
Type 2 diabetes mellitus is usually associated with high blood pressure, which is a risk factor for kidney disease. Aggressive blood pressure reduction is an important strategy to protect the kidney and reduce urinary protein which develops with kidney disease. This study will evaluate the effects of amlodipine/benazepril in reducing blood pressure and urinary protein in hypertensive subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate hypertension
* Type 2 diabetes mellitus
* Presence of protein in the urine (albuminuria)

Exclusion Criteria:

* Kidney disease not caused by diabetes or hypertension
* Renal artery stenosis
* Myocardial infarction or stroke within the last 6 months
* Type 1 diabetes mellitus
* Pregnant or lactating females
* Cancer within the last 5 years

Ages: 21 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 332 (Actual)
Dates: Start 2003-04; Primary Completion 2005-10 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the urine albumin/creatinine ratio after 52 weeks

SECONDARY OUTCOMES:
Percentage of patients who have progressed to diabetic kidney disease (urine albumin/creatinine ratio ≥ 300 µg/mg creatinine) after 52 weeks
Change from baseline in the ratio of urine albumin/creatinine ratio an estimate of kidney function after 52 weeks
Change from baseline in insulin resistance after 52 weeks
Change from baseline in urine albumin secretion after 52 weeks
Change from baseline in a marker of heart failure after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals